CLINICAL TRIAL: NCT03971955
Title: CharacterIzation of Adult Onset Autoimmune Diabetes
Acronym: CIAO
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1437923
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adult Onset Autoimmune Diabetes/Latent Autoimmune Diabetes
  Interventions: Other: Mixed Meal Test; Other: Dual Energy X-Ray Absorptiometry (DEXA); Procedure: Adipose Tissue Biopsy
- Type 2 Diabetes
  Interventions: Other: Mixed Meal Test; Other: Dual Energy X-Ray Absorptiometry (DEXA); Procedure: Adipose Tissue Biopsy
- Type 1 Diabetes
  Interventions: Other: Mixed Meal Test; Other: Dual Energy X-Ray Absorptiometry (DEXA); Procedure: Adipose Tissue Biopsy
- Healthy Normal Volunteers (HNV)
  Interventions: Other: Mixed Meal Test; Other: Dual Energy X-Ray Absorptiometry (DEXA); Procedure: Adipose Tissue Biopsy

INTERVENTIONS:
Other: Mixed Meal Test — a standard liquid mixed meal will be administered to the participant. The test meal with 1 kcal/ml and with the following caloric distribution Protein: 25%, Carbohydrate: 53%, Fat: 22% is given at a dose of 6 mL per kilogram body weight. Maximum dose is 360 mL and it will be ingested over 5 minutes. Blood samples will be taken 10 min prior to ingestion (t=-10), at baseline (t = 0), and at 15, 30, 60, 90, and 120 minutes.
Other: Dual Energy X-Ray Absorptiometry (DEXA) — DEXA Scans will be performed to obtain body composition measures (body fat and estimated muscle mass) using a General Electric (GE) Lunar iDXA whole-body scanner.
Procedure: Adipose Tissue Biopsy — The abdominal skin 6-10 cm lateral to the umbilicus will be cleansed with chlorhexidine. A sterile drape is placed, and the skin and adipose tissue will be anesthetized using Lidocaine. A 3-4 mm Mercedes Liposuction cannula will be inserted for aspiration of up to 2g of adipose tissue.

SUMMARY:
The purpose of the study is to identify new biomarkers of Adult Onset Autoimmune Diabetes (AOnAD).

ELIGIBILITY:
Inclusion Criteria:

Type 1 Diabetes (T1D)

* age 18-35 years
* age at diagnosis 13 to 30 years
* Body Mass Index (BMI) 25 to 35 kg/m2 with a stable body weight (±3 kg in the past 6 months)
* diagnosis of T1D according to American Diabetes Association (ADA) criteria continuously requiring insulin for survival (if in doubt, diagnosis can be confirmed by positivity of 2 or more IAAb* at time of diagnosis, at any time or at time of recruitment)
* diabetes diagnosis performed within the previous 5 years,
* requiring insulin continuously since diagnosis to prevent ketosis
* Fasting C-peptide levels < 0.3 nmol/l

Type 2 Diabetes (T2D)

* age 40-75 years
* age at diagnosis 40 to 70 years
* BMI 25 to 35 kg/m2 with a stable body weight (±3 kg in the past 6 months)
* diagnosis of diabetes according to ADA criteria
* Diabetes diagnosis performed within the previous 5 years
* Not requiring insulin
* Fasting C-peptide levels > 0.3 nmol/l

Adult Onset Autoimmune Diabetes/Latent Autoimmune Diabetes of Adults (AOnAD/LADA)

* age 40-75 years
* age at diagnosis 40 to 70 years
* BMI 25 to 35 kg/m2 with a stable body weight (±3 kg in the past 6 months)
* diagnosis of diabetes according to ADA criteria
* fasting C-peptide > 0.3 nmol/l
* positive for at least one islet autoantibody (IAAb* - at time of diagnosis, at any time or at time of recruitment)
* not requiring insulin or, if on insulin, treatment started at least 6 months after diagnosis

Healthy Normal Volunteers (HNV)

* age 40-75 years
* BMI 25 to 35 kg/m2 with a stable body weight (±3 kg in the past 6 months)
* No personal history of diabetes according to ADA criteria
* No history of diabetes in first degree relatives (FDRs)
* Fasting C-peptide levels > 0.3 nmol/l

  * IAAbs are Insulin AutoAntibodies (IAA), Thyrosine phosphatase IA-2 Antibodies (IA-2 Ab), Glutamic Acid Decarboxylase Antibodies (GAD Ab), Zinc Transporter 8 Antibodies (ZnT8 Ab), Islet Cell Antibodies (ICA).

Exclusion Criteria:

* For T2D participants: treatment with insulin or with thiazolidinediones (TZDs).
* For T1D and AOnAD/LADA participants: treatment with TZDs.
* Presence of unstable cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months, clinically significant abnormalities on EKG, presence of cardiac pacemaker, implanted cardiac defibrillator)
* Evidence of acute or chronic liver disease even if asymptomatic (AST or ALT >2.5 times the upper limit of normal)
* Kidney disease (creatinine >1.6 mg/dl or estimated GFR<60 ml/min)
* Triglycerides >500 mg/dl, LDL >200 mg/dl
* Uncontrolled hypertension (Blood Pressure BP>160 mmHg systolic or >100 mmHg diastolic)
* Recent important weight loss (>3 kg in 3 months)
* History of drug or alcohol abuse (> 3 drinks per day) within the last 5 years.
* History of cancer within the last 5 years (skin cancers, with the exception of melanoma, may be acceptable).
* History of organ transplant.
* History of bariatric surgery
* Bleeding or coagulation disorders requiring chronic use of blood thinners.
* Current treatment with blood thinners or antiplatelet medications that cannot be safely stopped for study procedures
* History of chronic pancreatitis or pancreatic surgery
* Acute or chronic infections
* History of HIV, active Hepatitis B or C, or Tuberculosis.
* Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women) or other chronic hematology disorders.
* Use of any medications known to influence glucose, fat and/or energy metabolism within the last 3 months (e.g., growth hormone therapy, glucocorticoids [steroids], etc.) other than the treatment for diabetes
* Thyroid dysfunction. Participants with a Thyroid Stimulating Hormone TSH > 10 µ IU or less than 0.4 µ IU are excluded. Participants on thyroid replacement medication or on antithyroid drugs may be enrolled providing they have been on a stable dose of medication for at least 6 weeks prior to screening and their TSH is within the range specified above.
* Severe asthma or chronic obstructive pulmonary disease
* Initiation or change in hormone replacement therapy within the past 3 months (including, but not limited to birth control or estrogen replacement therapy)
* Cushing's disease or syndrome
* Drugs that affect immune, weight or metabolic function, including but not limited to: oral corticosteroids, oral or injectable anti-obesity medications. Drugs for dyslipidemia (statins, ezetimibe, etc.) and a daily full strength or baby aspirin for atherosclerosis prevention will be allowed, provided patients have been on stable doses for at least 6 weeks prior to screening and that aspirin could be safely temporarily stopped for the study
* Weight >450 lbs. (This is Dual X-ray Absorptiometry (DEXA) table weight limit)
* Gastrointestinal disorders associated with malabsorption.
* Pregnant or nursing females or females less than 6 months postpartum from the scheduled date of collection.
* Had major surgery within 4 weeks prior to the pre-trial (screening) visit
* Participation in studies involving investigational drug(s) within 30 days prior to Screening Visit 1
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to Screening Visit
* Allergies to milk derived or soy derived products, lactose intolerance (due to the composition of the standard liquid meal that will be used for the test)
* Allergies and reactions to lidocaine.
* History of eating disorders
* Psychiatric disease prohibiting adherence to study protocol
* Unable to provide a reliable informed consent
* Presence of any condition that, in the opinion of the investigator and clinical team, compromises participant safety or data integrity or the participant's ability to complete study visits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an observational cross-sectional pilot study that will compare 4 groups of 10 participants each (5±1 of each gender per group) affected by AOnAD, T2D, T1D and Healthy Normal Volunteers (HNV). They will be characterized clinically and biochemically.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Blood collection | Screening Visit and Day 1
  A change in the levels of specific microRNAs (miRNA) isolated from circulating exosomes.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Casu, Principal Investigator — Study Principal Investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S13-S28. doi: 10.2337/dc19-S002. PMID 30559228
- [Background] Rogers MAM, Kim C, Banerjee T, Lee JM. Fluctuations in the incidence of type 1 diabetes in the United States from 2001 to 2015: a longitudinal study. BMC Med. 2017 Nov 8;15(1):199. doi: 10.1186/s12916-017-0958-6. PMID 29115947
- [Background] Thomas NJ, Jones SE, Weedon MN, Shields BM, Oram RA, Hattersley AT. Frequency and phenotype of type 1 diabetes in the first six decades of life: a cross-sectional, genetically stratified survival analysis from UK Biobank. Lancet Diabetes Endocrinol. 2018 Feb;6(2):122-129. doi: 10.1016/S2213-8587(17)30362-5. Epub 2017 Nov 30. PMID 29199115
- [Background] Thunander M, Petersson C, Jonzon K, Fornander J, Ossiansson B, Torn C, Edvardsson S, Landin-Olsson M. Incidence of type 1 and type 2 diabetes in adults and children in Kronoberg, Sweden. Diabetes Res Clin Pract. 2008 Nov;82(2):247-55. doi: 10.1016/j.diabres.2008.07.022. Epub 2008 Sep 18. PMID 18804305
- [Background] Thomas NJ, Lynam AL, Hill AV, Weedon MN, Shields BM, Oram RA, McDonald TJ, Hattersley AT, Jones AG. Type 1 diabetes defined by severe insulin deficiency occurs after 30 years of age and is commonly treated as type 2 diabetes. Diabetologia. 2019 Jul;62(7):1167-1172. doi: 10.1007/s00125-019-4863-8. Epub 2019 Apr 10. PMID 30969375
- [Background] Turner R, Stratton I, Horton V, Manley S, Zimmet P, Mackay IR, Shattock M, Bottazzo GF, Holman R. UKPDS 25: autoantibodies to islet-cell cytoplasm and glutamic acid decarboxylase for prediction of insulin requirement in type 2 diabetes. UK Prospective Diabetes Study Group. Lancet. 1997 Nov 1;350(9087):1288-93. doi: 10.1016/s0140-6736(97)03062-6. PMID 9357409
- [Background] Barinas-Mitchell E, Kuller LH, Pietropaolo S, Zhang YJ, Henderson T, Pietropaolo M. The prevalence of the 65-kilodalton isoform of glutamic acid decarboxylase autoantibodies by glucose tolerance status in elderly patients from the cardiovascular health study. J Clin Endocrinol Metab. 2006 Aug;91(8):2871-7. doi: 10.1210/jc.2005-2667. Epub 2006 May 23. PMID 16720660
- [Background] Insel RA, Dunne JL, Atkinson MA, Chiang JL, Dabelea D, Gottlieb PA, Greenbaum CJ, Herold KC, Krischer JP, Lernmark A, Ratner RE, Rewers MJ, Schatz DA, Skyler JS, Sosenko JM, Ziegler AG. Staging presymptomatic type 1 diabetes: a scientific statement of JDRF, the Endocrine Society, and the American Diabetes Association. Diabetes Care. 2015 Oct;38(10):1964-74. doi: 10.2337/dc15-1419. PMID 26404926
- [Background] Acevedo-Calado M, James EA, Morran MP, Pietropaolo SL, Ouyang Q, Arribas-Layton D, Songini M, Liguori M, Casu A, Auchus RJ, Huang S, Yu L, Michels A, Gianani R, Pietropaolo M. Identification of Unique Antigenic Determinants in the Amino Terminus of IA-2 (ICA512) in Childhood and Adult Autoimmune Diabetes: New Biomarker Development. Diabetes Care. 2017 Apr;40(4):561-568. doi: 10.2337/dc16-1527. Epub 2017 Feb 7. PMID 28174261
- [Background] Achenbach P, Hawa MI, Krause S, Lampasona V, Jerram ST, Williams AJK, Bonifacio E, Ziegler AG, Leslie RD; Action LADA consortium. Autoantibodies to N-terminally truncated GAD improve clinical phenotyping of individuals with adult-onset diabetes: Action LADA 12. Diabetologia. 2018 Jul;61(7):1644-1649. doi: 10.1007/s00125-018-4605-3. Epub 2018 Apr 4. PMID 29619531
- [Background] Brooks-Worrell BM, Boyko EJ, Palmer JP. Impact of islet autoimmunity on the progressive beta-cell functional decline in type 2 diabetes. Diabetes Care. 2014 Dec;37(12):3286-93. doi: 10.2337/dc14-0961. Epub 2014 Sep 19. PMID 25239783
- [Background] Buzzetti R, Zampetti S, Maddaloni E. Adult-onset autoimmune diabetes: current knowledge and implications for management. Nat Rev Endocrinol. 2017 Nov;13(11):674-686. doi: 10.1038/nrendo.2017.99. Epub 2017 Sep 8. PMID 28885622
- [Background] Hawa MI, Kolb H, Schloot N, Beyan H, Paschou SA, Buzzetti R, Mauricio D, De Leiva A, Yderstraede K, Beck-Neilsen H, Tuomilehto J, Sarti C, Thivolet C, Hadden D, Hunter S, Schernthaner G, Scherbaum WA, Williams R, Brophy S, Pozzilli P, Leslie RD; Action LADA consortium. Adult-onset autoimmune diabetes in Europe is prevalent with a broad clinical phenotype: Action LADA 7. Diabetes Care. 2013 Apr;36(4):908-13. doi: 10.2337/dc12-0931. Epub 2012 Dec 17. PMID 23248199
- [Background] Mishra R, Hodge KM, Cousminer DL, Leslie RD, Grant SFA. A Global Perspective of Latent Autoimmune Diabetes in Adults. Trends Endocrinol Metab. 2018 Sep;29(9):638-650. doi: 10.1016/j.tem.2018.07.001. Epub 2018 Jul 23. PMID 30041834
- [Background] Valadi H, Ekstrom K, Bossios A, Sjostrand M, Lee JJ, Lotvall JO. Exosome-mediated transfer of mRNAs and microRNAs is a novel mechanism of genetic exchange between cells. Nat Cell Biol. 2007 Jun;9(6):654-9. doi: 10.1038/ncb1596. Epub 2007 May 7. PMID 17486113
- See also: Translational Research Institute for Metabolism and Diabetes (TRI-MD) — https://www.adventhealth.com/research/translational-research-institute-metabolism-and-diabetes